CLINICAL TRIAL: NCT06898164
Title: The Influence of Axial Length on Visual Quality Following SMILE Surgery in Patients with High Myopia
Status: Completed | Type: Observational
Sponsor: yuhao shao (Other)
Collaborators: Shanghai 10th People's Hospital (Other)
Responsible Party: Sponsor-Investigator, yuhao shao, MD, Tongji University
Organization: Tongji University (Other)
Other Study IDs: 2025AL; YJXYS-B-009 (Other Grant/Funding Number: Shanghai 10th People's Hospital); 202240131 (Other Grant/Funding Number: Shanghai 10th People's Hospital)
Record Dates: First submitted 2025-03-13; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Visual Quality; Axial Length; High Myopia
Keywords: Axial length; High myopia; SMILE; Higher-order aberration; visual quality

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- AL < 26 mm: high myopic patients with axial lengths < 26 mm
  Interventions: Other: This study does not involve any interventions
- 26 mm ≤ AL < 27 mm: high myopic patients with 26 mm ≤ axial lengths < 27 mm
  Interventions: Other: This study does not involve any interventions
- AL ≥ 27 mm: high myopic patients with axial lengths ≥ 27 mm
  Interventions: Other: This study does not involve any interventions

INTERVENTIONS:
Other: This study does not involve any interventions — This study does not involve any interventions

SUMMARY:
This retrospective study aimed to investigate the subjective and objective visual outcomes following Small Incision Lenticule Extraction (SMILE) surgery in high myopic patients with varying axial lengths (AL).

DETAILED DESCRIPTION:
The study enrolled 113 highly myopic patients (202 eyes) who underwent SMILE surgery at Shanghai's Tenth People's Hospital. Patients were classified into three groups based on the axial length before surgery: Group A (AL < 26 mm, 62 eyes), Group B (26 mm ≤ AL < 27 mm, 88 eyes), and Group C (AL ≥ 27 mm, 52 eyes). Preoperative and postoperative evaluations included uncorrected distance visual acuity (UDVA), corrected distance visual acuity (CDVA), equivalent spherical error(SE), and corneal high order aberration. Subjective visual quality was assessed using the Quality of Vision (QoV) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* manifest refraction spherical equivalent refraction exceeding -6.00D;
* stable myopia for a duration of at least 2 years;
* corrected distance visual acuity of at least 20/25;
* annual myopic spherical equivalent increment less than - 0.50 D.

Exclusion Criteria:

* a history of moderate to severe dry eye as well as any ocular or systemic disease.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 113 high myopic patients (202 eyes) of Shanghai's Tenth People's Hospital were enroled in this prospective, non-randomized study conducted from July 2021 to September 2023.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Subjective visual quality | 12 months
  The quality of vision (QOV) questionnaire consists of (i) symptom frequency, (ii) severity, and (iii) bothersomeness for (a) glare, (b) halo, (c) starbursts, (d) hazy vision, (e) blurred vision, (f) distortion, (g) multiple images, (h) visual fluctuations, (i) difficulty focusing, and (j) difficulty judging distance or depth perception. Respondents use a scale of 0 to 3, where zero (0) denotes "none," one (1) "a little," two (2) "quite a bit," and three (3) "very much." Furthermore, on a scale from 0 to 10, patients were asked to provide Likert ratings for "daytime" and "nighttime" quality of vision (0 denoting the poorest vision, while 10 indicating the best vision)

SECONDARY OUTCOMES:
Refractive results | 12 months
  The uncorrected distance visual acuity (UDVA, logMAR), corrected distance visual acuity (CDVA, logMAR), subjective refraction (Diopter), and intraocular pressure (mmHg) were evaluated prior to and 1 year after SMILE.

OTHER OUTCOMES:
Ocular high-order aberrations | 12 months
  Corneal aberration measurements were performed using a Scheimpflug tomography system (Pentacam; Oculus GmbH, Wetzlar, Germany). Images of the highest quality (designated as OK) were selected for analysis. The coefficients for a standardized diameter of 8 mm were examined, followed by an assessment of the clinical significance of total higher-order aberrations (HOA, mm), spherical aberration (Z4, 0, mm), horizontal coma (Z3, 1, mm), vertical coma (Z3, -1, mm), horizontal trefoil (Z3, 3, mm), and oblique trefoil (Z3, -3, mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No